CLINICAL TRIAL: NCT01537302
Title: A Non-randomized Study of the Avinger Ocelot System Used to Cross Chronic Total Occlusions in the Superficial Femoral and Popliteal Arteries
Brief Title: Chronic Total Occlusion Crossing With the Ocelot System - CONNECT II
Acronym: CONNECTII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avinger, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVI OCT 10005
Record Dates: First submitted 2012-02-15; First posted 2012-02-23 (Estimated); Results first posted 2015-03-18 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Total Atherosclerotic Occlusion of Femoral Artery
Keywords: Chronic Total Occlusion; Optimal Coherence Tomography; Lumivascular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ocelot System (Experimental): CTO crossing in femoropopliteal arteries using the Ocelot System
  Interventions: Device: CTO crossing in femoropopliteal arteries CONNECT II

INTERVENTIONS:
Device: CTO crossing in femoropopliteal arteries CONNECT II — CTO crossing in femoropopliteal arteries using the Ocelot System
  Other Names: Chronic TOtal OcclusioN CrossiNg with thE OCelot SysTem II; CONNECT II

SUMMARY:
Evaluation of the safety and effectiveness of the Ocelot System to provide OCT-assisted orientation while simultaneously crossing totally occluded femoropopliteal arteries.

DETAILED DESCRIPTION:
The purpose of this clinical study is to evaluate the safety and effectiveness of the Ocelot System to provide OCT-assisted orientation while simultaneously crossing chronic total occlusions (CTOs) in femoropopliteal arteries. The Ocelot Catheter is a minimally invasive percutaneous device that is designed to traverse arterial occlusions through the use of spiral wedges contained in the distal tip of the device. The device is also equipped with an OCT (optical coherence tomography) imaging fiber that provides directional orientation and an intravascular view of the vessel wall and target lesion. The Ocelot Catheter is used in conjunction with standard endovascular devices and as an adjunct to fluoroscopic guidance.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to provide informed consent
* Patient is willing and able to comply with the study protocol
* Patient is > 18 years old
* Patient has peripheral arterial disease requiring revascularization as evidenced by CTA, MRA or angiography
* Patient has an occluded femoropopliteal artery that is 99-100% stenosed and is ≥ 1 cm and ≤ 30 cm in length by visual estimate
* Target vessel is ≥ 3.0 mm in diameter
* Patient has Rutherford Classification of 2-5
* Lesion is recalcitrant to guidewire crossing

Exclusion Criteria:

* Patient has a known sensitivity or allergy to contrast materials that cannot be adequately pre-treated
* Patient has a known sensitivity or allergy to aspirin, heparin or anti-platelet medications
* Patient is pregnant or lactating
* Patient has a co-existing disease or medical condition contraindicating percutaneous intervention
* Target vessel is severely calcified as evidenced by angiography
* Target lesion is in a bypass graft
* Target lesion is in a stent (i.e., in-stent restenosis)
* Patient has had a procedure on the target limb within 7 days
* Patient has had a procedure on the target limb within the past 30 days and is unstable
* Patient has a planned surgical or interventional procedure within 30 days after the study procedure
* Patient is simultaneously participating in an investigational device study for treatment of peripheral vascular disease
* Patient has a planned amputation of the target limb
* Patient has a history of bleeding diathesis, coagulopathy or will refuse blood transfusion in cases of emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Selmon, MD, Principal Investigator — Austin Heart Hospital; Arne Schwindt, MD, Principal Investigator — Muenster Hospital
Locations (17):
- United States (14):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Sutter Memorial, Sacramento, California
  - Cardiovascular Associates - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - St. Joseph's Hospital, Fort Wayne, Indiana
  - Detroit Medical Center, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - St. Dominic Hospital, Jackson, Mississippi
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Columbia University Medical Center, New York, New York
  - Jobst Vascular Center, Toledo, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Austin Heart, Austin, Texas
  - El Paso Cardiology Associates, El Paso, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
- Germany (2):
  - Leipzig Hospital, Leipzig
  - Muenster Hospital, Münster
- Mirano Hospital, Mirano, Italy

REFERENCES:
- See also: Avinger web site — http://www.avinger.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with CTO were approached to consider joining the study.
Period: Overall Study
Arm/Group | Ocelot System
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects.
Arm/Group | Ocelot System
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data unknown for 12 subjects.
  Participants
    Caucasian: number analyzed (Participants) | 88
    Caucasian | 64
    African American: number analyzed (Participants) | 88
    African American | 18
    Hispanic/Latino: number analyzed (Participants) | 88
    Hispanic/Latino | 3
    Asian: number analyzed (Participants) | 88
    Asian | 1
    American Indian: number analyzed (Participants) | 88
    American Indian | 0
    Native Hawaiian or Pacific Islander: number analyzed (Participants) | 88
    Native Hawaiian or Pacific Islander | 0
    Other: number analyzed (Participants) | 88
    Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 81
  Germany | 13
  Italy | 6
Rutherford [Count of Participants; unit: Participants]
  0 - Asymptomatic | 0
  1 - Mild Claudication | 0
  2 - Moderate Claudication | 13
  3 - Severe Claudication | 61
  4 - Ischemic Rest Pain | 20
  5 - Minor Tissue Loss | 6
  6 - Major Tissue Loss | 0
Ankle-Brachial Index [Count of Participants; unit: Participants] — Population: Data not obtained for 2 subjects.
  Participants
    ABI >1.3: Non-Compressible Vessels: number analyzed (Participants) | 98
    ABI >1.3: Non-Compressible Vessels | 0
    ABI ≥ 0.95: Normal: number analyzed (Participants) | 98
    ABI ≥ 0.95: Normal | 5
    ABI < 0.95: Peripheral Vascular Disease: number analyzed (Participants) | 98
    ABI < 0.95: Peripheral Vascular Disease | 47
    ABI < 0.6: Intermittent Claudication: number analyzed (Participants) | 98
    ABI < 0.6: Intermittent Claudication | 38
    ABI < 0.4: Chronic Limb Ischemia: number analyzed (Participants) | 98
    ABI < 0.4: Chronic Limb Ischemia | 8
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.7 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint
Description: No evidence of in-hospital MAEs, 30 day MAEs, clinically significant perforations, clinically significant embolizations or Grade C or greater dissections after Ocelot System CTO crossing confirmed by angiography.
Time Frame: Day 30
Population: Two subjects withdrew prior to 30-day follow-up.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Ocelot System
Number analyzed (Participants) | 98
Percent of participants | 2 [NA to 6.0] — This is a 95% one-sided confidence interval.

2. Primary Outcome: Primary Efficacy Endpoint
Description: Successful femoropopliteal CTO crossing using the Ocelot System as identified by guidewire placement in the distal true lumen confirmed by angiography.
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Ocelot System
Number analyzed (Participants) | 100
Participants | 97

3. Secondary Outcome: Procedural Success
Description: Successful delivery, crossing and retrieval of the investigational device in the absence of in-hospital MAEs, clinically significant perforations, clinically significant embolizations or Grade C or greater dissections.
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Ocelot System
Number analyzed (Participants) | 100
Participants | 95

4. Secondary Outcome: Technical Success
Description: Successful delivery, crossing and retrieval of the investigational device without the use of an assist device.
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Ocelot System
Number analyzed (Participants) | 100
Participants | 72

5. Secondary Outcome: Device Performance
Description: Device performance as assessed by Investigator's input by evaluating both performance of the device and quality of the OCT image as it relates to the ability to identify layered and non-layered structures and the ability of the directional marker bands to aid in orientation of the catheter while advancing through the CTO.
Time Frame: Day 0
Population: 'Catheter Performance Evaluation: Tip Deflection': Data was missing for one subject for this question.
  'OCT Performance Evaluation: Visualization of side branches': N/A in 9 subjects who did not have side branches visualized.
Measure: Count of Participants; unit: Participants
Arm/Group | Ocelot System
Number analyzed (Participants) | 100
Participants
  Catheter Performance Evaluation: Introduction into sheath: 5 - Excellent | 87
  Catheter Performance Evaluation: Introduction into sheath: 4 - Good | 13
  Catheter Performance Evaluation: Introduction into sheath: 3 - Acceptable | 0
  Catheter Performance Evaluation: Introduction into sheath: 2 - Poor | 0
  Catheter Performance Evaluation: Introduction into sheath: 1 - Unacceptable | 0
  Catheter Performance Evaluation: Catheter trackability: 5 - Excellent | 76
  Catheter Performance Evaluation: Catheter trackability: 4 - Good | 21
  Catheter Performance Evaluation: Catheter trackability: 3 - Acceptable | 3
  Catheter Performance Evaluation: Catheter trackability: 2 - Poor | 0
  Catheter Performance Evaluation: Catheter trackability: 1 - Unacceptable | 0
  Catheter Performance Evaluation: Catheter pushability: 5 - Excellent | 62
  Catheter Performance Evaluation: Catheter pushability: 4 - Good | 31
  Catheter Performance Evaluation: Catheter pushability: 3 - Acceptable | 6
  Catheter Performance Evaluation: Catheter pushability: 2 - Poor | 1
  Catheter Performance Evaluation: Catheter pushability: 1 - Unacceptable | 0
  Catheter Performance Evaluation: Tip Deflection: number analyzed (Participants) | 99
  Catheter Performance Evaluation: Tip Deflection: 5 - Excellent | 56
  Catheter Performance Evaluation: Tip Deflection: 4 - Good | 25
  Catheter Performance Evaluation: Tip Deflection: 3 - Acceptable | 18
  Catheter Performance Evaluation: Tip Deflection: 2 - Poor | 0
  Catheter Performance Evaluation: Tip Deflection: 1 - Unacceptable | 0
  Catheter Performance Evaluation: Ability to stay in true lumen: 5 - Excellent | 65
  Catheter Performance Evaluation: Ability to stay in true lumen: 4 - Good | 22
  Catheter Performance Evaluation: Ability to stay in true lumen: 3 - Acceptable | 10
  Catheter Performance Evaluation: Ability to stay in true lumen: 2 - Poor | 2
  Catheter Performance Evaluation: Ability to stay in true lumen: 1 - Unacceptable | 1
  Catheter Performance Evaluation: Visibility of radiopaque marker: 5 - Excellent | 82
  Catheter Performance Evaluation: Visibility of radiopaque marker: 4 - Good | 13
  Catheter Performance Evaluation: Visibility of radiopaque marker: 3 - Acceptable | 5
  Catheter Performance Evaluation: Visibility of radiopaque marker: 2 - Poor | 0
  Catheter Performance Evaluation: Visibility of radiopaque marker: 1 - Unacceptable | 0
  Catheter Performance Evaluation: Catheter tip visibility: 5 - Excellent | 84
  Catheter Performance Evaluation: Catheter tip visibility: 4 - Good | 13
  Catheter Performance Evaluation: Catheter tip visibility: 3 - Acceptable | 3
  Catheter Performance Evaluation: Catheter tip visibility: 2 - Poor | 0
  Catheter Performance Evaluation: Catheter tip visibility: 1 - Unacceptable | 0
  OCT Performance Evaluation: Clarity of images: 5 - Excellent | 63
  OCT Performance Evaluation: Clarity of images: 4 - Good | 31
  OCT Performance Evaluation: Clarity of images: 3 - Acceptable | 5
  OCT Performance Evaluation: Clarity of images: 2 - Poor | 0
  OCT Performance Evaluation: Clarity of images: 1 - Unacceptable | 1
  OCT Performance Evaluation: Visualization of layered structures: 5 - Excellent | 65
  OCT Performance Evaluation: Visualization of layered structures: 4 - Good | 22
  OCT Performance Evaluation: Visualization of layered structures: 3 - Acceptable | 11
  OCT Performance Evaluation: Visualization of layered structures: 2 - Poor | 1
  OCT Performance Evaluation: Visualization of layered structures: 1 - Unacceptable | 1
  OCT Performance Evaluation: Visualization of non-layered structures: 5 - Excellent | 63
  OCT Performance Evaluation: Visualization of non-layered structures: 4 - Good | 20
  OCT Performance Evaluation: Visualization of non-layered structures: 3 - Acceptable | 14
  OCT Performance Evaluation: Visualization of non-layered structures: 2 - Poor | 2
  OCT Performance Evaluation: Visualization of non-layered structures: 1 - Unacceptable | 1
  OCT Performance Evaluation: Visualization of side branches: number analyzed (Participants) | 91
  OCT Performance Evaluation: Visualization of side branches: 5 - Excellent | 60
  OCT Performance Evaluation: Visualization of side branches: 4 - Good | 24
  OCT Performance Evaluation: Visualization of side branches: 3 - Acceptable | 7
  OCT Performance Evaluation: Visualization of side branches: 2 - Poor | 0
  OCT Performance Evaluation: Visualization of side branches: 1 - Unacceptable | 0
  OCT Performance Evaluation: Flush adequately displaces blood for visualization: 5 - Excellent | 70
  OCT Performance Evaluation: Flush adequately displaces blood for visualization: 4 - Good | 28
  OCT Performance Evaluation: Flush adequately displaces blood for visualization: 3 - Acceptable | 2
  OCT Performance Evaluation: Flush adequately displaces blood for visualization: 2 - Poor | 0
  OCT Performance Evaluation: Flush adequately displaces blood for visualization: 1 - Unacceptable | 0
  OCT Performance Evaluation: Ability to orient using the middle marker: 5 - Excellent | 65
  OCT Performance Evaluation: Ability to orient using the middle marker: 4 - Good | 25
  OCT Performance Evaluation: Ability to orient using the middle marker: 3 - Acceptable | 10
  OCT Performance Evaluation: Ability to orient using the middle marker: 2 - Poor | 0
  OCT Performance Evaluation: Ability to orient using the middle marker: 1 - Unacceptable | 0
  OCT Performance Evaluation: Ability of OCT marker band to aid in catheter navigation: 5 - Excellent | 70
  OCT Performance Evaluation: Ability of OCT marker band to aid in catheter navigation: 4 - Good | 22
  OCT Performance Evaluation: Ability of OCT marker band to aid in catheter navigation: 3 - Acceptable | 7
  OCT Performance Evaluation: Ability of OCT marker band to aid in catheter navigation: 2 - Poor | 1
  OCT Performance Evaluation: Ability of OCT marker band to aid in catheter navigation: 1 - Unacceptable | 0

6. Secondary Outcome: Procedural Time
Description: Total time of the procedure from the insertion of the catheter to its removal following treatment of the CTO
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ocelot System
Number analyzed (Participants) | 100
minutes | 107.3 (57.5)

7. Secondary Outcome: Fluoroscopic Time
Description: Total time fluoroscopy was used during the procedure.
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ocelot System
Number analyzed (Participants) | 100
minutes | 38.6 (29.1)

8. Secondary Outcome: CTO Crossing Time
Description: Time required to cross the CTO during the procedure.
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ocelot System
Number analyzed (Participants) | 100
minutes | 32.9 (42.9)

9. Secondary Outcome: Use of Assist Devices
Description: Comparison of the crossing times for the Ocelot System alone versus the Ocelot System with assist devices.
Time Frame: Day 0
Population: Seventy-two participants in the 'CTO Crossing Time: Ocelot Alone'. Twenty-five participants in the 'CTO Crossing Time: Ocelot and assist devices'. Three subjects who did not have their CTO successfully crossed were excluded from calculation.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ocelot System
Number analyzed (Participants) | 100
minutes
  CTO Crossing Time: Ocelot Alone: number analyzed (Participants) | 72
  CTO Crossing Time: Ocelot Alone | 16.8 (18.4)
  CTO Crossing Time: Ocelot and assist devices: number analyzed (Participants) | 25
  CTO Crossing Time: Ocelot and assist devices | 79.1 (58.1)

10. Secondary Outcome: Contrast/Flush Volumes
Description: Contrast and flush volumes are presented
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Ocelot System
Number analyzed (Participants) | 100
ml
  Flush Volume (through Ocelot for visualization only) | 33.1 (57.9)
  Contrast Volume (used for entire procedure) | 223.0 (144.7)
  Contrast Volume (procedure start through CTO crossing) | 124.5 (100.3)

ADVERSE EVENTS:
Time Frame: Day 0 through Day 30
Arm/Group | Ocelot System
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 26/100
Other Adverse Events (participants affected / at risk) | 25/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocelot System (N=100)
AV Fistula (Injury, poisoning and procedural complications) | 1 (1)
Vessel Dissection, Grade C or greater (Injury, poisoning and procedural complications) | 1 (1)
Vessel Dissection, Grade A or B (Injury, poisoning and procedural complications) | 3 (3)
Bruising or hemorrhage at procedural access site (Vascular disorders) | 3 (4)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Thrombosis (Vascular disorders) | 3 (3)
Pain, new or worsening (Vascular disorders) | 3 (3)
Infection (Infections and infestations) | 3 (3)
Pseudoaneurysm (Vascular disorders) | 3 (3)
Bleeding (other than access site) (Vascular disorders) | 1 (1)
Hypotension, sustained (Vascular disorders) | 3 (3)
Perforation requiring intervention (Injury, poisoning and procedural complications) | 3 (3)
Shortness of breath (Cardiac disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Perforation, not requiring intervention (Injury, poisoning and procedural complications) | 1 (1)
Acute COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
limb ischemia (Vascular disorders) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Allergic reaction to contrast medium (Immune system disorders) | 1 (1)
Altered mental state (Psychiatric disorders) | 1 (1)
Leg ulcerations (Vascular disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Intractable nausea/vomiting (Gastrointestinal disorders) | 1 (1)
Lethargy (General disorders) | 1 (1)
Uncontrolled hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocelot System (N=100)
Bruising or hemorrhage at procedural access site (Vascular disorders) | 9 (9)
Swelling (Vascular disorders) | 5 (5)
Bleeding, other than access site (Vascular disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Dysphagia (Nervous system disorders) | 1 (1)
Nausea/Vomiting (General disorders) | 4 (4)
Pain, new or worsening (General disorders) | 3 (3)
Perforation not requiring intervention (Injury, poisoning and procedural complications) | 2 (2)
Pseudoaneurysm (Vascular disorders) | 1 (1)
Vessel dissection, Grade A or B (Vascular disorders) | 5 (5)
Vessel dissection, Grade C or greater (Vascular disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
AV fistula (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the earliest of (a)publication of results, (b)receipt of notice stating that Study has been terminated or (c)18 months after completion or termination, Institution/Investigator (IN) shall have right to publish information & data collected or produced, provided that drafts are provided to Sponsor (SP) at least 60 days prior to the first submission. SP shall comment within 45 days. IN shall delay publication/presentation to enable SP to secure patent or other proprietary protection.